CLINICAL TRIAL: NCT01464957
Title: Skin Cancer Prevention in a Pediatric Population
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Kaiser Permanente (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 96-0014; R01CA074592 (NIH)
Record Dates: First submitted 2011-08-14; First posted 2011-11-04 (Estimated); Last update posted 2013-01-25 (Estimated); Status verified 2013-01

CONDITIONS: Skin Cancer
Keywords: skin cancer prevention; precaution adoption process model; semi-tailored newsletter; pediatric; behavioral intervention
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Newsletter intervention (Experimental): Semi-tailored newsletter intervention for parents and children
  Interventions: Behavioral: Semi-tailored newsletter
- Usual care (No Intervention): No newsletter intervention

INTERVENTIONS:
Behavioral: Semi-tailored newsletter — Delivered over 3 consecutive years, in the spring
  Other Names: Semi-tailored newsletter intervention; for parents and children
  Arms: Newsletter intervention

SUMMARY:
Skin cancer risk is largely determined by sun exposure during childhood. This study determines the effectiveness of a mailed intervention designed to increase sun protection for children age 6-9 years old. The intervention includes newsletters for parents that include risk information tailored to each child. Also included are sun protection resources such as a swim shirt, a sun hat, and sunscreen. Participants receive the intervention over 3 consecutive years, and data collection includes telephone interviews and skin exams. The study hypothesis is that receipt of the intervention will result in improved sun protection of the child.

DETAILED DESCRIPTION:
About 1 in 90 American children born in the late 1990's will develop malignant melanoma in their lifetimes. Sun exposure in childhood appears to be the most important preventable risk factor for this disease. This project will develop a tailored, risk-based, written intervention, which will be mailed to parents of children age 6-9 years in the spring of each year. The tailored intervention will utilize the Precaution Adoption Process Model, which has a primary focus on risk perception and suggests that there are seven stages leading to sustained health behavior change. The effectiveness of the intervention will be tested using a randomized controlled trail involving 1000 children recruited from health care facilities and community locations at age 5-6 years and followed for 3 years using telephone interviews to assess sun protection behaviors and skin exams to observe changes in melanocytic nevi, freckling, and tanning.

ELIGIBILITY:
Inclusion Criteria:

* Child born in 1998, has resided in the Denver, Colorado area

Exclusion Criteria:

* Parents unable to respond to telephone survey; child has disabling condition

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 867 (Actual)
Dates: Start 2003-11; Primary Completion 2007-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
sun protection behavior scale | change from baseline over 4 years
  Parent report through telephone interview

SECONDARY OUTCOMES:
Nevus counts | Change from baseline over 4 years
  Health care provider skin examination of nevi by size and body location

CONTACTS AND LOCATIONS:
Overall Officials: Lori A Crane, PhD, MPH, Principal Investigator — University of Colorado, Denver; Joseph Morelli, MD, Principal Investigator — University of Colorado, Denver; Stefan T Morelli, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Derived] Crane LA, Asdigian NL, Baron AE, Aalborg J, Marcus AC, Mokrohisky ST, Byers TE, Dellavalle RP, Morelli JG. Mailed intervention to promote sun protection of children: a randomized controlled trial. Am J Prev Med. 2012 Oct;43(4):399-410. doi: 10.1016/j.amepre.2012.06.022. PMID 22992358